CLINICAL TRIAL: NCT06759129
Title: RomSi (Rompiendo El Silencio) Mobile Health Intervention to Enhance Suicide Prevention by Reducing Stigma and Increasing Literacy: Protocol for a Cross-Over Randomized Controlled Trial
Brief Title: RomSi: Mobile Health Intervention to Enhance Suicide Prevention by Reducing Stigma and Increasing Literacy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Rosa M. Baños Rivera, Full Professor of Psycology, University of Valencia
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: VH9FA3L6BJ015JSE
Record Dates: First submitted 2024-12-10; First posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-12

CONDITIONS: Suicidal Ideation and Behavior; Suicide
Keywords: Suicide Prevention; Stigma; Suicide Literacy; Help Seeking; Randomized Controlled Trial
MeSH Terms: conditions — Suicidal Ideation; Behavior; Suicide; Suicide Prevention; Social Stigma | interventions — 1-(diethylaminopropyl)-4-phenylpiperazine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate-use (Experimental): Participants will use the mobile application starting immediately after the baseline assessment (T0) for approximately 14 days or until they complete the app.
  Interventions: Behavioral: Immediate-use of a mobile health application until completion
- Delayed use (Active Comparator): Participants will start using the application 14 days after the baseline assessment (T0) and immediately after the T1 assessment.
  Interventions: Behavioral: Delayed use of a mobile health application until completion

INTERVENTIONS:
Behavioral: Immediate-use of a mobile health application until completion — Participants will use the RomSi app for approximately 14 days, completing all scheduled activities. Throughout the intervention, they will respond to ecological momentary assessments (EMA) designed to evaluate stigma, help-seeking intentions, and suicidal ideation.
  The activities within the app will include interactive games aimed at fostering empathy and emotional understanding. Participants will also have continuous access to specialized help contacts to ensure their well-being during the study.
  The protocol involves two groups that will receive tailored information based on their specific needs:
  1. Individuals with low suicidal ideation and/or self-stigma, who will engage in activities focused on reducing personal stigma.
  2. Individuals experiencing suicide bereavement, who will receive support tailored to address their loss and foster resilience.
  A follow-up will be carried out one month and three months after the end of the intervention.
  Other Names: iApp
  Arms: Immediate-use
Behavioral: Delayed use of a mobile health application until completion — Participants assigned to the dApp group (delayed use) will not have access to the RomSi app during the first two weeks of the study. During this period, they will complete ecological momentary assessments (EMA) to evaluate stigma, help-seeking intentions, and suicidal ideation, without engaging in the intervention activities associated with the app.
  After completing this initial control phase, participants in the dAPP group will begin using the RomSi app, following the same protocol as the iAPP group. This includes interactive activities, such as games designed to foster empathy and understanding, along with continuous access to specialized help contacts.
  This crossover design allows for the immediate effects of the intervention to be compared between groups, while also evaluating changes in pre- and post-intervention measures across both conditions.
  A follow-up will be carried out one month and three months after the end of the intervention.
  Other Names: dApp
  Arms: Delayed use

SUMMARY:
Suicide is one of the leading causes of death in Spain, representing a public health crisis that requires urgent and effective solutions. The stigma surrounding suicide prevents many at-risk individuals from seeking help, worsening the problem. Addressing this stigma is essential to implement more effective and accessible prevention strategies. This study aims to design and evaluate an innovative mobile health intervention to reduce stigma and encourage help-seeking behaviours in the general population. While the intervention targets the general population, two specific groups will access specialized and tailored content: individuals with low suicidal ideation and family members or close friends of people who have died by suicide. Ecological Momentary Assessments (EMA) will collect real-time data and evaluate the intervention's impact. The study will employ a randomised controlled trial (RCT) with a crossover design, with participants randomly assigned to immediate or delayed use conditions. The intervention's effectiveness and usability will be assessed at four key points through quantitative analyses and qualitative interviews. We hypothesise that the intervention will improve suicide literacy, reduce suicide-related stigma, increase help-seeking behaviours, and demonstrate high usability and acceptability.

DETAILED DESCRIPTION:
Despite advances in suicide prevention research, implementation faces significant challenges. One major obstacle is stigma, which discourages many at-risk individuals from seeking help and hinders public awareness and societal commitment to addressing this issue openly and responsibly.

Public stigma includes negative beliefs, such as perceiving individuals with suicidal thoughts as "weak" or "selfish." This stigma can be internalized by those experiencing suicidal ideation or behaviour, negatively affecting their self-esteem and increasing their distress and isolation due to fear of rejection. Furthermore, family members and friends who have lost a loved one to suicide also face stigma, complicating their grieving process and increasing their risk of depression.

This context highlights the need for effective interventions to reduce stigma, encourage help-seeking, and provide support for both at-risk individuals and their loved ones.

The goal of this study is to develop and validate a mobile application called RomSi ("Rompiendo el silencio" in Spanish; Breaking the Silence), designed to improve knowledge about suicide, reduce associated stigma, and promote help-seeking behaviours. The app incorporates four intervention approaches that have proven effective in other mental health stigma reduction programs:

1. Psychoeducation,
2. Interpersonal contact,
3. Cognitive flexibility, and
4. Values-based work.

Additionally, the app will leverage innovative tools like Ecological Momentary Assessment (EMA) to collect real-time data and personalize the intervention to each participant's needs. Gamification elements will also be used to enhance motivation and engagement throughout the intervention.

To evaluate the effectiveness of RomSi, a randomized controlled trial (RCT) with a crossover design will be conducted. Participants will be randomly assigned to one of two groups:

* iApp: Immediate use of the app.
* dApp: Delayed use (waitlist control).

The randomization process will use a computer-generated sequence, concealed from researchers until group assignment, and stratified based on stigma levels toward suicide.

Evaluations will occur at five key time points:

* T0 (pre-intervention): Initial questionnaires.
* T1 (post-intervention): After app completion (iApp) or after 14 days of waiting (dApp).
* T2: Follow-up 14 days after T1.
* T3: Follow-up 1 month.
* T4: Follow-up 3 months.

The iApp group will begin using the app immediately after T0 and will have 14 days to complete it, though they may proceed at their own pace. The dApp group will act as a waitlist control, starting the app after completing T1 and following the same evaluation schedule.

During the intervention, EMA will be used to measure stigma levels daily, while suicidal ideation and help-seeking behaviors will be assessed at T0, at 7 days, and at the end of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years old or older.
* Have a cell phone with internet access during the intervention and follow-up periods.
* Be able to speak, understand, and read in Spanish.

Exclusion Criteria:

* Presence of high suicidal ideation (measured during screening, with a score above 20 on the total SIDAS scale or between 7 and 10 on the item assessing suicide attempts).
* Presence of high social desirability bias (measured during screening, with a score of 14 or higher on the MC-SDS scale).
* Altered mental status that impedes the ability to provide informed consent or assent (e.g., acute psychosis, intoxication, or mania).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 214 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Suicide public stigma | Assessments will be conducted at enrollment, immediately after app completion (14 days after enrollment for the iApp group or at the end of the control phase for the dApp group), and at one-month and three-month follow-ups.
  Public stigma will be assessed using the Spanish version of the Stigma of Suicide Scale - Short Form (SOSS-SF). This scale includes 16 adjectives that prototypically describe a person who has died by suicide. It is designed for use with the general population and identifies three distinct factors: (1) Stigma (e.g., pathetic), (2) glorification/Normalization (e.g., brave), and (3) isolation/Depression (e.g., lonely). Each item is rated on a 5-point Likert scale, where higher scores indicate stronger agreement with the adjective as a representation of a prototypical suicidal person.
Suicide literacy | Assessments will be conducted at enrollment, immediately after app completion (14 days after enrollment for the iApp group or at the end of the control phase for the dApp group), and at one-month and three-month follow-ups.
  The Literacy of Suicide Scale - Short Form (LOSS-SF) will be used to assess levels of suicide-related knowledge. The Spanish validation comprises 10 items divided into four domains: (1) signs and symptoms, (2) causes or nature, (3) risk factors, and (4) treatment and prevention. Responses are provided on a three-point scale ("true," "false," "don't know"). Each correct response is awarded one point, with higher scores indicating greater literacy about suicide.
Intention to seek help | Assessments will be conducted at enrollment, immediately after app completion (14 days after enrollment for the iApp group or at the end of the control phase for the dApp group), and at one-month and three-month follow-ups.
  The General Help-Seeking Questionnaire (GHSQ) measures the intention to seek help from various sources. Participants rate 10 items regarding their likelihood of seeking help on a 7-point scale ranging from 1 (extremely unlikely) to 7 (extremely likely) for 10 different help sources. The questionnaire provides an overall score and two subscale scores: formal help sources and informal help sources, with higher scores indicating greater help-seeking intention.
EMA questionnaire protocol | Public stigma will be assessed daily during the 14-day intervention period. Help-seeking intention and suicidal ideation will be assessed at four specific time points throughout the intervention.
  Participants will be assessed daily using ecological momentary assessments (EMA) to evaluate public stigma toward suicide, suicidal ideation, and help-seeking intention. Public stigma will be measured using words derived from the literature and the previously mentioned SOSS questionnaire. help-seeking intention will be assessed with a specific item, while suicidal ideation will be evaluated using the Spanish version of the Suicidal Ideation Attributes Scale (SIDAS).

SECONDARY OUTCOMES:
Personal suicide stigma | This measure will only be implemented for participants with low or moderate suicidal ideation. Assessments will be conducted at enrollment, immediately after app completion (14 days after enrollment for the iApp group or at the end of the control phase f
  The Personal Suicide Stigma Questionnaire (PSSQ) will be used to assess individuals' perceptions of social responses to their experiences with suicidal behaviour. It comprises 16 items rated on a 5-point Likert scale (1 = never to 5 = very often) and includes three subscales: Rejection, Minimization, and Self-Blame. The total score ranges from 16 to 80, with higher scores indicating greater experiences of suicide-related stigma.
Suicide grief experience | This measure will only be implemented for participants who indicate bereavement as a consequence of suicide in the screening. Assessments will be conducted at enrollment, immediately after app completion (14 days after enrollment for the iApp group or at
  The Grief Experience Questionnaire (GEQ) will be used to assess feelings arising from the experience of suicide among individuals close to the deceased. The scale consists of 55 items that measure the frequency of specific reactions experienced during the two years following the loss, rated on a 5-point Likert scale (1 = never to 5 = almost always). The items are distributed across 11 subscales.
Stigma by association towards suicide. | Assessments will be conducted at enrollment, immediately after app completion (14 days after enrollment for the iApp group or at the end of the control phase for the dApp group), and at one-month and three-month follow-ups.
  The Stigma of Suicide and Suicide Survivor Scale (STOSASS) will be used to assess perceived stigma toward suicide and suicide survivors. The tool consists of two subscales: one for stigma toward suicide and another for stigma toward survivors, each comprising 13 items rated on a 4-point scale (1 to 4). The total score is calculated as the average of the 13-item scores, with higher total scores indicating greater perceived stigma.

OTHER OUTCOMES:
Depressive symptoms | Assessments will be conducted at enrollment, immediately after app completion (14 days after enrollment for the iApp group or at the end of the control phase for the dApp group), and at one-month and three-month follow-ups.
  The Patient Health Questionnaire-9 (PHQ-9) will be administered. This is a nine-item scale based on the DSM-IV diagnostic criteria for major depression. Responses are recorded on a 4-point Likert scale reflecting the frequency of symptoms over the past two weeks, ranging from 0 ("Never") to 3 ("Nearly every day"). Additionally, the final question assesses the level of difficulty these issues have caused, using a 4-point Likert scale from 1 ("Not difficult at all") to 4 ("Extremely difficult"). Higher scores indicate greater severity of depressive symptoms.
Anxious symptoms | Assessments will be conducted at enrollment, immediately after app completion (14 days after enrollment for the iApp group or at the end of the control phase for the dApp group), and at one-month and three-month follow-ups.
  The Generalized Anxiety Disorder 7-item scale (GAD-7) will be administered to assess the presence and severity of generalized anxiety disorder. Participants will respond to 7 items regarding the frequency of their experiences over the past two weeks, using a scale ranging from 0 ("Not at all") to 3 ("Nearly every day").
Suicidal ideation | Assessments will be conducted at enrollment, immediately after app completion (14 days after enrollment for the iApp group or at the end of the control phase for the dApp group), and at one-month and three-month follow-ups.
  The severity of suicidal ideation will be assessed using the Suicidal Ideation Attributes Scale (SIDAS), which consists of 5 items. These items evaluate the frequency of suicidal thoughts (item 1), the ability to control them (item 2), proximity to a suicide attempt (item 3), associated distress (item 4), and interference with daily activities (item 5) over the past month. Responses are recorded on an 11-point Likert scale, with scores above 21 indicating a high risk of suicidal behavior.
Expectations and opinions on the intervention | Immediately before and after the intervention
  Expectations and Opinion of Treatment Scales consist of two 5-item scales that provide a subjective measure of participants' expectations and opinions about the treatment. Items are rated on a 0-to-10 Likert scale, with higher scores indicating more positive expectations or opinions.
Usability | Immediately after the intervention
  The System Usability Scale (SUS) is a 10-item questionnaire that evaluates the usability of a technological application.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No